# Manual of Operations and Procedures

## **Project CLEAR Changing Lives by Eradicating Antibiotic Resistance**

Funded by: Agency for Healthcare Research and Quality

Principal Investigator: Susan S. Huang, MD, MPH

## **Table of Contents**

| Introduction | |
|----------------------------------------------------------------|----|
| 1. List of Abbreviations and Definition of Terms | 5 |
| 2. Forms and Binders | 7 |
| 2.1 Forms | 7 |
| 2.2 Binders and Files. | 8 |
| 2.3 Logs | 8 |
| 3. Key Personnel | |
| 4. Participating Centers | 10 |
| 5. Identification Numbers | 11 |
| 6. Assessing Eligibility for Recruitment | 11 |
| 7. Inclusion/Exclusion Criteria | |
| 8. Informed Consent Process | |
| 9. Recruitment/Enrollment Study Visit | |
| 9.1 Stratification | |
| 9.2 Randomization | |
| 9.3 Participant Education | |
| 9.4 Surveys | |
| 9.5 Body Site Swabbing | |
| 9.5.1 Swabbing Technique: Nasal | |
| 9.5.2 Swabbing Technique: Throat | |
| 9.5.3 Swabbing Technique: Inguinal Region and Axilla | |
| 9.5.4 Swabbing Technique: Open Wounds | |
| 9.6 Study Intervention | |
| 9.7 Scheduling Next Visit | |
| 9.8 Scheduling Bi-Monthly Phone Calls | |
| 9.9 Physician Letters | |
| 9.10 Product Start Date/Study Start Date | |
| 10. Central Office Reference Guide | |
| 10.1 Daily Tasks | |
| 10.2 Day-Specific Tasks | |
| 10.3 Recurring Tasks | |
| 10.4 Morning Routine | |
| 10.5 Randomization | |
| 10.6 Patient Tracking Log. | |
| 10.7 Scheduling Appointments | |
| 10.8 Assigning Appointments | 28 |
| 10.9 Rescheduling and Cancelling Appointments | 28 |
| 10.10 Disenrolling Patients | |
| 10.11 Adverse Events | |
| 10.12 Medical Visit Reporting | |
| 10.13 Scanned Consents/Releases | |
| 10.14 Creating Consent/Recruitment and Follow-Up Visit Packets | |
| 10.15 PCP Letters | 34 |

## Project CLEAR MOP Version 1.3 April 7, 2011

| 10.16 | 5 Exit Survey | 34 |
|--------|-----------------------------------------------|----|
| 10.17 | Reports | 34 |
| 10.18 | Shipping | 35 |
| 10.19 | P End of Day Laboratory Email | 35 |
| | Study Products | |
| 11. | Follow-Up Participant Tracking and Scheduling | 36 |
| 11.1 | Patient Contact | 36 |
| 11.2 | Calendars | 37 |
| 11.3 | Call Lists | 37 |
| | Patient Phone Calls | |
| 11 | .4.1 Initial Post-Discharge Phone Call | 37 |
| | .4.2 Reminder Calls | |
| | .4.3 Product Review/Orientation Calls | |
| | Study Helpline | |
| 12. I | Bi-Monthly Phone Calls | 39 |
| | Follow-up Study Visits | |
| | Participant Education | |
| 13.2 | Interviews | 41 |
| | Adverse Events | |
| | Medical Events | |
| | Body Site Swabbing | |
| | Scheduling Next Visit | |
| | Update Contact Information | |
| | Participant Payments | |
| | Off Site Follow-Up Visits | |
| | .9.1 Home Visit Procedures | |
| | Adverse Event Reporting | |
| | Obtaining Medical Records | |
| | Data Entry | |
| | Ordering Supplies | |
| | Enrollment Reports | |
| 19. \$ | Specimen Delivery and Order Entry | 48 |

## Introduction

This Manual of Operations and Procedures (MOP) will be used to standardize study procedures for the clinical trial, "Project CLEAR - Changing Lives by Eradicating Antibiotic Resistance". Study personnel are to refer to this document when conducting all study procedures. If there are further questions or clarification is needed please call/email the Senior Project Coordinator Supervisor

#### 1. List of Abbreviations and Definition of Terms

Abbreviation

Arm of the study:

E: Education Group

D: Decolonization and Education Group

CHG: Chlorhexidine gluconate. The active antiseptic ingredient in the Hibiclens body wash and Perioguard mouthwash.

ICF: Informed Consent Form. A form that must be signed by subjects documenting their willing participation in the study. The ICF explains the objectives, design, risks, and benefits of the study including compensation for participating.

ID: Identification. As in identification number for a person or center.

Study ID numbers associated with ethnicity/location:

1,000's and 6,000's NN: Non-Hispanic/Not long term care facility

2,000's HN: Hispanic/Not long term care facility

3,000's NL: Non-Hispanic/Long term care facility

4,000's HL: Hispanic/Long term care facility

IRB: Institutional Review Board. A faculty committee charged with reviewing and approving the use of human subjects in all research projects to ensure that the safety and welfare of subjects are protected.

LTC: Long-term care facility. A facility such as a nursing home, skilled nursing facility, or rehabilitation center that subjects may be discharged to, rather than house/apartment/condo/townhouse.

MRSA: Methicillin Resistant Staphylococcus aureus.

MSSA: Methicillin Sensitive Staphylococcus aureus.

PHI: Protected Health Information.

S. aureus: Staphylococcus aureus.

Specimen Sources:

NA Nares

TH Throat

SK Skin (axilla/groin)

WD Wound (if applicable for not all patients will have wounds)

UCI: University of California, Irvine. The primary investigative team site.

UCI-CO: UCI Central Office. The call center to be contacted when randomizing a patient.

VTOC: Vision Tree Optimal Care. Web-based database application used for tracking and maintaining study data for Project CLEAR.

#### Visit Numbers:

R0 Recruitment/Enrollment visit

V1 Month 1 visit

V2 Month 3 visit

V3 Month 6 visit

V4 Month 9 visit

PT: Participant

6

#### 2. Forms and Binders

#### **2.1 Forms**

All forms for subjects will be available in English and Spanish.

#### ICF:

1. Adult Informed Consent Form + PHI Authorization

#### Questionnaires:

- 1. Participant Screening Form
- 2. Participant Identifier Enrollment Contact Information
- 3. Participant Enrollment Survey
- 4. Participant Identifier Follow up Contact Information
- 5. Participant Follow up Survey (Education)
- 6. Participant Follow up Survey (Decolonization)
- 7. Adverse Event Reporting Form
- 8. Medical Visit Reporting Form
- 9. Trial Exit Survey

#### Other:

- 1. Field Checklist
- 2. Initial Hospital Visit
- 3. Consented Patient (Identifier)
- 4. Facilities
- 5. Travel
- 6. Staff Directory
- 7. IRB
- 8. Q & A
- 9. Study Procedures Checklist
- 10. Directions for forms and surveys
- 11. Shipping Specimen Tracking Form
- 13. Educational Handouts
- 14. Specimen Labels
- 15. Calendar
- 16. Missed Appointments Letter
- 17. Study Product

#### 2.2 Binders and Files

<u>Recruitment Log File Folder</u> (Contains: Recruitment, Consent, and Count Logs for each recruitment center)

<u>Subject File</u> (Contains: ICF, medical information release form, contact sheet, all questionnaires, adverse event forms and medical event forms. Each subject will have one binder)

<u>Subject Study Binder</u> (Contains: study and visit information, MRSA Education and Decolonization

<u>Lab Results Binder</u> (Contains: Colonization lab results)

## **2.3 Logs**

<u>Central Office Enrollment Log</u> (List of all randomized and enrolled participants from the various participating centers, including the participant's name, study ID, recruiter, hospital, discharge date, and first follow-up visit)

<u>Central Office Lab Count Log</u> (List of the number of specimen swabs with corresponding Study ID numbers collected daily from each recruiter and hospital and sent to the UCI Microbiology Lab for processing)

<u>Recruitment Log</u> (List of eligible MRSA positive patients from each participating center—see Figure 6.1)

<u>Consent Log</u> (List of enrolled patients from each individual participating center to be kept at the facility—See Figure 6.2)

<u>Count Log</u> (Count of potential participants who enrolled, declined, or were missed at each participating center)

## 3. Key Personnel

#### **Faculty - UCI:**

Susan Huang – Principal Investigator Steven Park – Co-investigator Dan Gillen - Statistician

#### **Study Staff - UCI:**

Raveena Singh – Sr. Clinical Research Coordinator, Supervisor Adrijana Gombosev – Senior Clinical Research Coordinator Victor Quan – Senior Clinical Research Coordinator Suzie Hong – Clinical Research Coordinator

Eric Cui – Assistant Clinical Research Coordinator

Diane Kim – Assistant Clinical Research Coordinator

Cameron Lee – Assistant Clinical Research Coordinator

Syma Rashid – Assistant Clinical Research Coordinator

Courtney Reynolds – MD, PhD candidate

Chenghua (Mick) Cao – Programmer Analyst

Jiayi He – Programmer Analyst

Thomas Tjoa – Programmer Analyst

Qixin (Bay) Wang – Programmer Analyst

#### **Recruiters – UCI (Assistant Clinical Research Coordinator):**

Stephanie Arredondo-Glacet

Elizabeth Arreola

Donald Bayley

Claudia Cervantes

Heather Clayton

Nhi Dam

Tabitha Dutciuc

Lauren Heim

Brian Lewis

Andrea Marcantonio

Lisa "Angie" McErlain

Belinda Prado

Ivonne Turner

**Emily Wawro** 

#### **Central Office - UCI (Assistant Clinical Research Coordinator):**

Nelly Beltran

Sandra Ibarra

Maureen Schroeder

#### Central Office Coordinators (Medical Records Request and Redaction):

Jennifer Do – Assistant Clinical Research Coordinator

Phillip Duffy – Assistant Clinical Research Coordinator

Marlene Estevez – Assistant Clinical Research Coordinator

Usme Kushbu – Assistant Clinical Research Coordinator

Jennifer Lequieu – Assistant Clinical Research Coordinator

Nicole Mohaier – Assistant Clinical Research Coordinator

Jennifer Nam – Assistant Clinical Research Coordinator

Hanna Owens – Assistant Clinical Research Coordinator

Lauren Akahoshi – Junior Specialist

Deborah Prunean – Junior Specialist

Justin Chang – Research Assistant

#### **Institute for Clinical and Translational Science (ICTS):**

Angela Mendoza – Front Office Barbara Bodenhoefer – ICTS Nurse Diane Capobianco – ICTS Nurse Melanie Meton – ICTS Nurse

#### **UC Irvine Microbiology Lab**

Kaye Evans – Microbiology CLS Supervisor Maria Mejia – Microbiology Clinical Laboratory Scientist Cynthia Toyoshima – Microbiology Clinical Laboratory Scientist

#### **Harbor-UCLA:**

Loren Miller – Co-Investigator James McKinnell – Co-Investigator Michael Bolaris - Co-Investigator Samantha Eells – Program Coordinator Jenna Alcaron – Study Coordinator Isabel Alegria – Study Coordinator Ramiro Correa – Study Coordinator Nathalia Cressey – Study Coordinator Margarita Flores – Study Coordinator Ann Nguyen – Study Coordinator Katy Precaido – Study Coordinator Sean Prendergast – Study Coordinator Diana Romero – Study Coordinator Aubrianne Rose – Study Coordinator Grace Tagudar - Study Coordinator Raul Macias-Gil – Lab/Medical Records Review Jun Zozobrado – Medical Records Requests

#### **Ventura County Medical Center:**

Gail Simpson – Co-Investigator Stefan Boghossian – Student Intern/Recruiter

## 4. Participating Centers

#### **Hospitals:**

Downey Regional Medical Center Fountain Valley Regional Hospital Harbor-UCLA Medical Center Hoag Memorial Hospital Presbyterian Little Company of Mary, San Pedro Little Company of Mary, Torrance Long Beach Memorial Medical Center Mission Hospital – Laguna Beach
Mission Hospital – Mission Viejo
Orange Coast Memorial Medical Center
Saddleback Memorial Medical Center – Laguna Hills
Saddleback Memorial Medical Center – San Clemente
St. Jude Medical Center
St. Mary Medical Center
Torrance Memorial Medical Center
UC Irvine Medical Center
Ventura County Medical Center

#### **Nursing Homes:**

Chapman Care Center
Country Villa Plaza Convalescent Center
Covington Care Center
Pacific Haven Healthcare
Regents Point - Windcrest
Royale Healthcare Center
Villa Elena Healthcare

#### 5. Identification Numbers

Subjects ID numbers are: D or E followed by a four-digit number – NN, HN, HL, NL

D represents patients randomized to the decolonization arm

E represents patients randomized to the education arm

NN represents patients enrolled in the non-Hispanic, non-long-term care facility stratum (see stratification section 9.1)

HN represents patients enrolled in the Hispanic, non-long-term care facility stratum

HL represents patients enrolled in the Hispanic, long-term care facility stratum

NL represents patients enrolled in the non-Hispanic, long-term care facility stratum

Subject ID numbers and Arms (D or E) will be assigned using the next sequential assignment within the appropriate strata (NH, HN, HL, NL) per statistician-created randomization file as pulled from the randomization block by the UCI Central Office (UCI-CO)

## 6. Assessing Eligibility for Recruitment

Each medical center may have a slightly different preferred method of identifying MRSA positive cultures and eligible individual screening. The information below applies in general to our participating centers.

#### Positive MRSA cultures:

Infection prevention and control personnel at each site will notify study personnel about the eligible inpatients who have a positive MRSA culture (either clinical culture or nasal swab) by providing a line list of positive cultures from the hospital microbiology lab.

#### **Contacting Potential Patients:**

All patients with a MRSA positive culture will be recorded in the Recruitment Log (Figure 6.1). For all patients with a positive culture that are not enrolled, the reason why the patient is not approached or enrolled will be recorded according to the following matrix:

| CODE | STATUS |
|---|---|
| MISS | Missed opportunity for recruitment, patient not approached for recruitment |
| D1 | Declined, minimal to no pitch |
| D2 | Declined, moderate pitch |
| D3 | Declined, full pitch |
| CONSENT | Patient consented |

Figure 6.1. Recruitment Log



If an eligible patient is still hospitalized, the study coordinator will approach the patient in the hospital. Recruiters will leave either a note or the consent form in the medical record. Prior to approaching the patient, the recruiter will speak with the patient's nurse (as the patient may not have been told they have MRSA yet). Once the patient's nurse approves, the recruiter will then speak with the patient in their room to determine whether they wish to participate in the study. Subjects that agree to participate will be consented at this time. Patients who are unsure or unavailable will be recorded in the recruitment log by the coordinator so that the patient can be approached again at a later time. For patients who need additional time to think about the trial, a brochure will be left with them with information about the trial. Trial declinations will also be recorded in the Recruitment Log.

When approaching a patient in person, the coordinator should have all current versions of the consent form and PHI form with them. Study binders and/or study product will be provided to the patient by the coordinator following consent and randomization and will be kept in a temporary storage location at the facility until the patient is ready to be discharged.

Eligible patients that agree to participate will be consented and recorded in the Consent Log (Figure 6.2).

Eligible patients who were hospitalized, but have now been discharged: If the patient's treating MD during the hospitalization gives permission to contact them, the study coordinator will call the patient at the phone number listed on the hospital chart to approach the patient and use the treating MD's name to explain how we are reaching out to them. If the eligible patient does not answer, the study coordinators will leave a message stating that the patient is eligible for a research study. In the message, study coordinators will not mention that the eligible patient had an MRSA infection or colonization. If the patient verbally agrees to participate, the patient must be consented and complete their baseline visit at the clinic within 30 days of hospital discharge. If the potential patient is unable to come into the clinic, study coordinators may schedule a home visit or nursing home visit with the patient.

Eligible patients who are being discharged to a LTC facility: The study coordinators will call all facilities to make them aware that a patient has enrolled in the study. For LTC facilities not already engaged in study participation, study coordinators will call the facility that the eligible patient will be discharged to and assess the willingness of the center to participate. Study coordinators will also be available to visit the facility per patient needs, introduce Project CLEAR, and provide instructions on study protocol, *e.g.*, bathing instructions.

Eligible patients who call central office due to the media campaign: Patients who call the 800 number because they have seen or heard one of the study advertisements will speak to study coordinators over the phone to determine eligibility. Patients deemed to be meet inclusion criteria will have a visit scheduled for enrollment. Patients must provide documentation of a hospitalization and a MRSA positive culture within 30 days of hospitalization in order to be enrolled.

Figure 6.2. Consent Log

| CONSENT LOG | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| # | ACRC<br>Initials | Last Name | First Name | Study ID | Room &<br>Ward | Contact<br>Sheet<br>Y/N | Enroll<br>Survey<br>Y/N | Give<br>Prod<br>Y/N | V1<br>Date<br>Y/N | DC<br>Date | DC Location<br>Type, Name<br>& City |
| 1 | | | | | | | | | | | |
| 2 | | | | | | | | | | | |
| 3 | | | | | | | | | | | |
| 4 | | | | | | | | | | | |
| 5 | | | | | | | | | | | |
| 6 | | | | | | | | | | | |
| 7 | | | | | | | | | | | |
| 8 | | | | | | | | | | | |
| 9 | | | | | | | | | | | |
| 10 | | | | | | | | | | | |

#### 7. Inclusion/Exclusion Criteria

The Inclusion and Exclusion Criteria Checklist should be reviewed with the patient to determine the patient's eligibility for the study.

#### **Inclusion Criteria**:

- 1) 18 years of age or older
- 2) Have a recent hospitalization (within the past 30 days)
- 3) Have an MRSA positive culture identified by microbiology laboratory
- 4) Able to provide their consent to participate or have a surrogate provide consent
- 5) Must be able to bathe, shower, or have this task performed daily by a caregiver (if applicable)

#### **Exclusion Criteria**:

- 1) The subject is allergic to mupirocin
- 2) The subject is allergic to chlorhexidine
- 3) Subject is receiving end-of-life hospice measures

#### 8. Informed Consent Process

The UCI and LA BioMed institutional Standard Operating Procedures will be utilized as a guide for consenting patients. Inpatients will be consented in a private or semi-private setting (usually their hospital room). Eligible patients who are contacted over the phone will be consented at the research clinic, home, or long-term care facility.

If the patient is more comfortable speaking in Spanish, a Spanish-speaking study coordinator should be contacted to approach the patient.

#### 9. Recruitment/Enrollment Study Visit

The baseline enrollment visit must occur either in the hospital before discharge or within 30 days of hospital discharge. Items required for the baseline visit include: enrollment survey, contact survey, required swabs, study product, and review of the arm-specific toolkit binder.

#### 9.1 Stratification

Once a patient has been consented, each subject will be classified into one of four groups:

- 1) Non-Hispanic ethnicity and long-term care facility (NL)
- 2) Hispanic ethnicity and long-term care facility (HL)
- 3) Non-Hispanic ethnicity and non-long-term care facility (NN)
- 4) Hispanic ethnicity and non-long-term care facility (HN)

Hispanic ethnicity is based upon self-report (or surrogate report) and long-term care facility refers to the subject being discharged to a nursing home. Assisted living does not qualify for long term care stratification. The ethnicity and facility information will be required by the UCI-CO at randomization. Study coordinators should collect this information prior to enrollment.

#### 9.2 Randomization

Subjects will be randomized by calling the UCI Central Office (CO) at will be answered between the hours of 8:00 and 17:30. Study coordinators must call CO as soon as the subject completes all enrollment and informed consent processes. Study coordinators must have the subject's name, gender, ethnicity, and LTC status. The project coordinator at UCI-CO will utilize the stratified randomization charts developed by statistician and provide the next available assignment number and arm in chronological order. The study coordinator will inform the patient of their randomization assignment and proceed to the next steps. For after-hours enrollment, please call the Project Coordinator Supervisor.

## 9.3 Participant Education

Each participant will be provided with an educational binder in his or her preferred language (English or Spanish). Subjects randomized to the Education Arm will receive an education only binder. Subjects randomized to the Decolonization Arm will receive the same education material as part of the decolonization binder. The study coordinator will review the binder with the participant. It is important to note that study coordinators cannot provide information other than what is specified in the binder. Study coordinators cannot extend specific medical advice to anyone. If participants have further questions they should be instructed to contact their physician.

## 9.4 Surveys

Surveys will be administered in-person by study coordinators. If the participant does not know or remember the answer, remind the participant to answer as best they can and move on the next question. Patients are encouraged to answer all questions and skip questions only when necessary. The survey interview should take no more than 20 minutes.

## 9.5 Body Site Swabbing

All participants will be swabbed using a BBL<sup>TM</sup> CultureSwab<sup>TM</sup> for *S. aureus* colonization at four body sites: the bilateral nares, throat, groin and axilla as a combined swab, as well as any wounds that the patient might have. The body swabs should be sent to the central lab within 24 hours for processing.

## 9.5.1 Swabbing Technique: Nasal

The study coordinator will place a sterile culture swab into the anterior nares of the participant as shown in Figure 9.5.1.



Figure 9.5.1: Depicts nasal chambers, nares (pear-shaped apertures) and vestibule. The culture swab is shown inserted through the anterior nares (nostril vestibule) to make contact with nasal membrane.

- A. Label sample by placing the pre-printed label on the outside of the sleeved device.
- B. Use "nares swab" label sticker.
- C. Write subject ID number, date/time collected on the label with a permanent marker (Sharpie or similar).
- D. Remove the protective sleeve of the culture swab exposing the shaft and rayon fiber bud. Only touch the outer hub of the swab without contacting the swab or shaft.
- E. Insert swab into sterile transport tube to moisten the swab. If the swab accidentally touches anything that is non-sterile (e.g. outside of transport tube), discard and begin again.
- F. Tell patient the swab is being moistened with sterile fluid. Tell them you will only go as far "as someone would put their finger in."
- G. Insert tip of swab 1-2 cm into nares. Insert the sterile culture swab into right anterior nares into the nostril vestibule toward the apex of the nose to make contact with the nasal mucous membrane (see Figure 1)
- H. Gently rotate the culture swab for two full turns while in contact with the nasal membrane.
- I. Gently withdraw the culture swab from right nares.
- J. With the same culture swab, gently repeat insertion and rotation on the left side
- K. Carefully re-sleeve the culture swab.
- L. Bury tip of culture swab in gel at bottom of tube.

#### 9.5.2 Swabbing Technique: Throat

The study coordinator will place a sterile culture swab into throat (tonsil area) of the participant as shown in Figure 9.5.2.



Figure 9.5.2: Depicts the throat and tonsillar area. The culture swab is shown touching (swabbing) the tonsil.

- A. Explain to patient what you are about to do.
- B. Label sample by placing the pre-printed label on the outside of the sleeved device.
- C. Use "throat swab" label sticker.
- D. Write subject ID, date/time collected on the label with a permanent marker.
- E. Remove the protective sleeve of culture swab exposing the shaft and rayon fiber bud.
- F. Only touch the outer hub of the swab without contacting the swab or shaft.
- G. Insert swab into transport tube to moisten the swab. If the swab accidentally touches anything that is non-sterile (e.g. outside of transport tube), discard and begin again.
- H. Tell patient the swab is being moistened with sterile fluid.
- I. Have patient tilt head back, breathe deeply open mouth wide and have them say "Ah". This serves to lift the uvula and aids in reducing the gag reflex.
- J. Use tongue depressor to gently depress the tongue, if necessary (consider moistening the tongue depressor with tap water if the participant gags).
- K. Every effort should be made to avoid touching the swabs to the tongue, teeth, roof of the mouth or the inside of the cheeks.
- L. Carefully but firmly rub the swabs over:
  - a. Both of the tonsils (or tonsilar crypts if tonsils have been removed).
  - b. Posterior pharynx (back of throat).
- M. Remove swabs carefully from the mouth, again avoid touching the swabs to the tongue, teeth, roof of the mouth or the inside of the cheeks.
- N. Carefully re-sleeve the culture swab.
- O. Bury tip of culture swab in gel at bottom of tube.

## 9.5.3 Swabbing Technique: Inguinal Region and Axilla

- A. Explain to patient what you are about to do.
- B. Label sample by placing the pre-printed label on the outside of the sleeved device.
- C. Use "inguinal/axilla swab" label sticker.
- D. Write subject ID, date/time collected on the label with a permanent marker.
- E. Remove the protective sleeve of culture swab exposing the shaft and rayon fiber bud.
- F. Only touch the outer hub of the swab without contacting the swab or shaft.
- G. Insert swab into transport tube to moisten the swab. If the swab accidentally touches anything that is non-sterile (e.g. outside of transport tube), discard and begin again.
- H. Tell patient the swab is being moistened with sterile fluid.
- I. Put sterile culture swab at bottom Right armpit (See Figure 9.3).
- J. Swab with upwards motion from bottom to top of R armpit fold.
- K. While moving culture swab, upwards, simultaneously rotate swab at least two complete turns.
- L. With same culture swab, repeat technique on the Left armpit fold.
- M. With same culture swab, use a similar technique to swab the R groin.
- N. With same culture swab, use a similar technique to swab the L groin.
- O. Carefully re-sleeve the culture swab.
- P. Bury tip of culture swab in gel at bottom of tube.



Figure 9.5.3: Depicts the left and right inguinal folds that should be swabbed

#### 9.5.4 Swabbing Technique: Open Wounds

Only wounds that are accessible should be swabbed. Do not disturb wounds that are inaccessible (occlusive dressing) or have a wound vac on.

- A. Explain to patient what you are about to do.
- B. Label sample by placing the pre-printed label on the outside of the sleeved device.
- C. Use "wound swab" label sticker.
- D. Write subject ID, date/time collected on the label with a permanent marker.
- E. Remove the protective sleeve of the culture swab exposing the shaft and rayon fiber bud.
- F. Only touch the outer hub of the swab without contacting the swab or shaft.
- G. Insert swab into transport tube to moisten the swab. If the swab accidentally touches anything that is non-sterile (e.g. outside of transport tube), discard and begin again.
- H. Tell patient the swab is being moistened with sterile fluid.
- I. Roll the swab over the wound, attempt to sample any drainage
- J. Carefully re-sleeve the culture swab.
- K. Bury tip of culture swab in gel at bottom of tube.

## **9.6 Study Intervention**

Subjects may be given their arm-specific toolkit binder and/or study materials (decolonization products) under four different scenarios:

- 1) On the day of enrollment The study coordinator may provide the toolkit binder to the study participant at the time of enrollment once randomized to the respective Education or Decolonization arm.
- 2) At hospital discharge In an effort to not lose study materials during a prolonged hospital stay, study coordinators may return on the day of discharge to provide the subject with their toolkit binder and study materials. Some medical centers may deliver the study materials (toolkit binder or decolonization products) at discharge via the pharmacy.
- 3) After discharge If a subject is discharged without receiving their toolkit binder or decolonization products or if they misplace their study products during their hospital stay the study material will be mailed or delivered to their home.
- 4) In clinic/home visit/nursing facility If a subject is recruited and enrolled outside of a hospital setting (at home, at the study clinic, or at a nursing home), the study coordinators will provide the toolkit binder and study materials at the time and place of enrollment. The toolkits will be reviewed in full with each participant at the time of receipt.

The study toolkit will contain:

Decolonization Group:

- 1) Study product (nasal mupirocin, CHG body wash (Hibiclens) and mouth wash)
- 2) Calendar cling
- 3) Copy of the consent form
- 4) Adverse Event form
- 5) Medical Visit Reporting form
- 6) Arm-specific educational binder
- 7) Appointment reminder card

#### **Education Group:**

- 1) Copy of the consent form
- 2) Adverse Event form
- 3) Medical Visit Reporting form
- 4) Arm-specific educational binder
- 5) Appointment reminder card

The recruiter is responsible for assigning the decolonization patients to the Plan A or Plan B schedule based upon week of start. The assignment to Plan A or Plan B is based on the first day of the initial five day decolonization cycle post discharge.

Once the patient is informed of the schedule that he or she follow, the study coordinator will remind the participant to start bathing for five consecutive days after being discharged from the hospital. The study coordinator will explain to the patient that after five day post discharge bathing regimen, they will follow the assigned calendar Plan A or Plan B calendar schedule. The

study coordinator will also remind the participant that UCI CO will call to remind them of the decolonization bathing schedule prior to the five-day CHG bathing cycle. The study coordinator will also instruct the participant to add an additional day to the end of their bathing regimen if a day is skipped during their assigned bathing cycle. In the event that the participant misses two or more days of the decolonization bathing cycle, they will have to restart the regimen.

The patient will be told that all of the products that they receive are used to reduce bacteria. The study coordinator will then instruct the study participant on how to use each study product and remind that the decolonization products must all be used together:

Hibiclens: "This chlorhexidine soap is a body wash/shampoo that needs to be used anytime you shower when you are scheduled to be on your five-day regimen. It is intended to substitute your body wash, shampoo and facial cleanser. Do not get product into eyes or ear canal. Also, it is very important to keep the product on your skin for two minutes while out of the water stream or reapply on the skin twice while out of the water stream for a total of two minutes Also, it is very important to keep the product on your skin for two minutes while out of the water stream before rinsing. The two minutes is approximately the time to soap up twice out of the water stream before rinsing." The study coordinator will also provide and demonstrate how to use the two-minute waterproof sand timer. Bactroban Nasal: "This mupirocin ointment is a prescription nasal ointment that needs to be used twice a day, in the morning and in the evening, when you are scheduled to be on your five-day regimen cycle. You will use half a tube for each nostril and dispose the empty tube into the container that is provided."

PerioGard: "This bottle is a chlorhexidine oral rinse that needs to be used twice a day, morning and evening, when you are scheduled to be on your five-day regimen cycle. You need to make sure you brush your teeth prior to swishing the oral rinse in your mouth for 30 seconds. Do not rinse your mouth with water after using this product. Also, make sure not to eat for at least a half an hour after using the oral rinse."

The study coordinator will remind the patient that if they have any study-related questions, they may call the toll-free study telephone number where the UCI Central Office will answer any questions regarding the study or study products.

## 9.7 Scheduling Next Visit

The study recruiter will make every effort to schedule the one month follow-up visit while conducting the enrollment visit if possible. If the participants cannot schedule the follow up visit at the time of enrollment, they will be provided with an appointment reminder card with a date that the visit should occur (approximately 30 days after discharge). The central office will call the participant two weeks prior to the time when the one-month follow-up should occur in order to schedule a fixed follow up appointment day, time, and location. See protocol for visit schedule.

## 9.8 Scheduling Bi-Monthly Phone Calls

Bi-monthly reminder phone calls should be scheduled the Friday before the start date of the intervention week. Central Office staff will reference the Study Contact Sheet to verify the best times to call based on indicated availability

## 9.9 Physician Letters

Participants are informed that, shortly after study enrollment, a notification letter will be sent to the participant's primary physician as well as be placed in their chart during hospitalization for the inpatient attending physician to see. The letter informs the physician of their patient's participation Project CLEAR and informs the physician of the study group that their patient has been randomized to (i.e. Education or Decolonization). The UCI Central Office will be responsible for sending letters to all study participant's physicians on their behalf.

#### 9.10 Product Start Date/Study Start Date

The product start date vs. trial start date, they are the same date, labeled differently in Vision Tree and databases. Study start date (aka. "Trial entry date" in our analytics dataset for Dan Gillen) is termed "product start date" in Vision Tree surveys and was used to capture study start date for both Decolonization and Education subjects.

Admit Date (Hosp) – Admit date of the recruitment hospitalization Trial Start Date – Generally the date of discharge or the date of enrollment if enrollment was performed post-discharge.

#### 10. Central Office Reference Guide

Below is a reference guide describing the daily and weekly tasks of central office coordinators for Project CLEAR.

#### 10.1 Daily Tasks

- Randomize patients and update tracking log, Recruitment Progress Report will be sent out daily to study investigators and senior project coordinator supervisor
- Create and send out swab collection email
- Call patients for next day's appointments

## 10.2 Day-Specific Tasks

- Monday: Bathing Regimen Cycle Reminder Calls
- Tuesday: Assign follow-up visits two weeks out (for example, on week one, schedule visits for week three). Scheduling should occur at least two weeks prior to the visit.
- Wednesday: Prepare UCI Missed Visit Names report, call patients who have missed visits (in person or for Trial Exit Report) and send out Missed Appointment Letter Thursday: Based on Trial Exit Report, schedule courtesy visits for potential Loss to Follow Up patients for coming week
- Friday: Prepare and send out Trial Exit Report, Prepare Monday Bathing Regimen Reminder Call List

#### 10.3 Recurring Tasks

Note: These do not have to be done on any particular day of the week, but must be done regularly each week, so as to remain current.

- Create participant consent and follow up visit folders.
- Scan patient consents and medical release forms. Call patients needing exit surveys from the UCI List.
- Create swab bags containing.
  - Specimen Sheets Biohazard Bags and Lab Requisition forms (carbon copy duplicates)
  - Swabs
- Create and send out Primary Care Physician letters.
- Maintain supply of compensation forms for recruiters.

## 10.4 Morning Routine

- 1. Obtain "enrollment log" & "specimen log" from locked cabinet.
- 2. Check voice mailbox to listen to voice messages left from after-hours calls
- 3. Locate "Patient Tracking Log" and update with current date

#### 10.5 Randomization

1. Log in VTOC with username & password. Click on "New Patient"



2. In VTOC enter the below information. Indicate if PT is *Hispanic* and if PT is going to a *nursing home* (Check Yes or No for both)



- 3. Provide recruiter with new Study ID #
- 4. Schedule V1 with recruiter or provide available days/times for patient's location
  - a. For more information, see **Scheduling Appointments** (page 6)
- 5. Ask the recruiter for the swab count and fill out Lab Count Log (note recruiter may need to give swab count to you later in the day)
- 6. On paper Enrollment Log, write in recruitment date, recruiter initials, hospital name, patient first and last name, and note swab count in margin.
- 7. Edit the Contact Sheet in VTOC and select the appropriate recruiter's name in the Recruiter Name pull down. Enter Visit One Date.
- 8. Under "initial recruitment" click new record to create a new "Participant Screening Form" ADD today's date and verify inclusion criteria

- 9. Click <u>new record</u> to create "participant enrollment survey"- ADD today's date ONLY. Note that Today's Date indicates the Consent Date, not the date data entry was done.
  - a. If patient was consented POST DISCHARGE, add name of original hospital in hospital field. Ex: Hospital: UCI PD (LBM)
- 10. Input new participant information into Patient Tracking Log
- 11. Text Senior Project Coordinator Supervisor information: 1-(recruiter(initials)\(hospital initials)\)
  - Example: 1-IT\UCI

## 10.6 Patient Tracking Log

Study patient information is entered into the "tracking log" and applicable information will be transferred over to VTOC.

The following information can be found on the "tracking log"

- 1. Patient ID & initials- An asterisk (\*) will be placed after the ID # for Spanish speakers.
- 1. Decolonization Plan (differentiated by color: (A-Green or B-Orange)
- 2. Discharge date
- 3. Recruiter Initials
- 4. Notes: used for comments regarding any communication with the patient (optional)

**IMPORTANT NOTES** are in **RED** (Ex: Do NOT call, email pref., Spanish speaking etc).

- 5. Initial bathing dates (1<sup>st</sup> & 5<sup>th</sup> day)
- 6. Date that the primary care provider was mailed notification
- 7. Consent scanned (Y for Yes)
- 8. Clinic visit dates, time & location
- 9. Date exit survey completed
- 10. Bathing cycle dates (1<sup>st</sup>day)

## 10.7 Scheduling Appointments

**ALL** appointments should be entered in the following locations:

- 1. VTOC:
  - a. Contact Sheet's Visit Field: Visit One, Visit Two, Visit Three, Visit Four
  - b. Communication Log: "HOME VISIT (V#) Date @ Time; Assigned to [Staff Name]."
- 2. Patient Tracking Log:

Date, time, location and geographic area (ie: 8/30/13 @12PM Home4)

3. ENDMRSA calendar – Sample set up:



- a. Categorize (Colors listed below) and Invite Attendees
- 4. Enrollment Log (V1 only)

#### **ENDMRSA Calendar Color Codes:**

- 1. Blue= Home, NH, hospital
- 2. Red= ALL cancellations /no shows
- 3. Green= Melanie (Wednesdays) appointments
- 4. Light green=Product review/product drop-off/courtesy visit
- 5. Light blue= Recruitment visits (post-discharge)
- 6. Yellow = Institute for Clinical and Translational Science (ICTS) Irvine/Orange

#### Visit Scheduling by Area

- 1. Institute for Clinical and Translational Science (ICTS) Nurse Visits
  - a. Monday, Friday ICTS Orange
  - b. Tuesday, Thursday ICTS Irvine
  - c. Wednesday ICTS nurse visits Area 3, 4 and 5 (double check address, must be within 15 miles of ICTS Irvine)
- 2. Home Visits
  - a. As possible, the coordinators are to group Area Visits together and in descending order of distance
    - i. Geographically distant visits should be scheduled earlier in the morning if possible, so that recruiters can go farthest distance in the morning, and work their way back in the afternoon
- 3. Home Visits (Spanish)
  - a. Schedule when PT is available, but try to group area appointments together (i.e. if staff is in Area 4 on Thursday, try to schedule Area 4 visits around that appointment)

#### **ICTS Appointments**

- 1. Create New Appointment on End MRSA Calendar
- 2. Subject: PT ID number (with asterisk if patient is Spanish speaking)
- 3. Location: ICTS (Orange or Irvine); Visit Number (V1, V2, V3, V4)
- 4. Select Time
- 5. Message: Patient name and marital status
- 6. Invite Attendees: End MRSA, ICTS Scheduling Coordinator and ICTS Nurse.
- 7. Categorize as Yellow
- 8. Note Appointment in Patient Tracking Log

#### **Home/NH Appointments**

- 1. Create New Appointment on End MRSA Calendar
- 2. Subject: PT ID number (with asterisk if patient is Spanish speaking)
- 3. Location: Home(Area Number) / NH(Area Number); Visit Number (V1, V2, V3, V4)
- 4. Select Time
- 5. Message: Patient name
- 6. Invite Attendees: End MRSA
  - a. If scheduling home visit for Melanie on Wednesday, also invite: ICTS Scheduling Coordinator and ICTS Nurse
- 7. Categorize as Blue
- 8. Note Appointment in Patient Tracking Log

**Remote Visits** – Rare. Should only occur when patient has moved out of the area (e.g. another state), but is still participating. Relates to collecting swabs from patients out of the coverage area

- 1. Call patient before their next visit due date and set up delivery and return of swabs for FedEx labels.
- 2. Create Visit Packet to overnight to participant
  - a. Study Visit Packet Contents:

Decolonization participants receive products for V1 and V2 (V3 and V4 do not receive study product) in addition to items listed below

- i. Visit Survey Questionnaire with a "CONFIDENTIAL" envelope (this will need to be picked up from UCIMC Micro Lab)
- ii. Swab bag (label the stickers and study paperwork with Visit #, Study ID, swab collection site (Na, Thr, Sk, Wd) and date that the patient is to complete swabbing
- b. Compensation
  - i. Subject Compensation Form

- Fill out the following: Date Paid, Cash (with corresponding visit amount), Amount Paid, Home Visit CASH Sign Out (your signature) and PT signs "Paid To" column Overnight to PT
- ii. Compensation (wait until signed compensation is received)
  - \$ in small envelope labeled and sealed "VISIT [#] COMPENSATION FOR: \_\_\_\_\_

iii. FedEx Package

#### **10.8** Assigning Appointments

- There will be one primary study coordinator for home visits
  - Try to make sure that there is as little duplication of area assignments as possible (if one study coordinator is conducting an appointment in Area 4, ensure that a second study coordinator does not have to drive there as well).
    - Note: study coordinators will be assigned to area visits that are closest to their geographical location (home)
- All Spanish appointments will be assigned to a Spanish speaking study coordinator. Senior Project Coordinator Supervisor will also receive an invitation as an FYI)
- Post-discharge R0 Enrollment Visit appointments should be scheduled according to the regular home visit schedule and study coordinators assigned to the closest geographical area

Note: R0 Enrollment Visit appointments will typically require a full hour and should be scheduled accordingly and take driving time into consideration as well

## 10.9 Rescheduling and Cancelling Appointments

- 1. If an appointment is CANCELLED- change category to RED, indicate CANCELLED next to Study ID, add today's date w/ notes in comments section.
- 2. If an appointment is RESCHEDULED-keep same color category (unless it needs to be changed), update date and time, add current date and notes in comments section, and resend a new appointment invitation.
  - i. Note: Keep original appointment on the calendar & create a new calendar appointment if study coordinator drove to destination but the appointment had to be rescheduled for any reasons.
- 3. Inform ICTS Scheduling Coordinator of any ICTS cancellations or reschedules by editing existing calendar invite.

- a. If it is a last minute cancellation or reschedule, make sure to also call the ICTS Appointment Center.
- 4. Save new date & time to: tracking log, contact sheet & communication log (VTOC).

#### **10.10 Disenrolling Patients**

Patients are considered to be an "early" exit/disenrollment if they exit the study due to death, active disenrollment, or confirmed lost to follow up.

#### **Active Disenrollment**:

- 1. If a patient expresses that they cannot participate in the study, the study coordinators will document reasons for withdrawing participation, attempt to address concerns and encourage continued participation, if possible. During the disenrollment interview, the coordinator is to attempt to gather outcomes data from the patient (they will ask if the participant has been re-hospitalized or has visited a clinic for a possible infection).
- 2. Fill out a Medical Visit Reporting Form if applicable
- 3. If they are adamant about dropping, notify the Senior Project Coordinator Supervisor via email and cc: the patient's recruiter and End MRSA email account.
  - a. In the email, the participant's ID # will be included in the subject line and a brief summary of the situation will be described in the body of the email.
- 4. A summary of the disenrollment event will also be recorded in the VTOC Communication Log.
- 5. After the Senior Project Coordinator Supervisor has followed up with patient, the patient will be added to the Trial Exit Report.
- 6. The patient will also be added to the "Physician Follow Up" Spreadsheet (Non-Participant List tab) for follow-up discussions and documented decisions regarding trial exit.
- 7. The VTOC Enrollment survey will also be updated
  - a. Complete Change of Enrollment Status section
    - i. Click YES
    - ii. Enter Date Disenrolled
    - iii. Set Reason Disenrolled to DECLINE
    - iv. Select the appropriate value for Reason Declined and give description under Notes.
      - 1. IMPORTANT: If no known outcome data is obtained during this time, use last date patient provided outcome data (Ex: RO, V1).

## Project CLEAR Participant Enrollment Survey



- 8. Update Patient Tracking Log
  - a. Highlight patient entry in red
  - b. Note "Active disenrollment" and "Supervisor notified" in comments section

#### Death:

- 1. If study staff is informed that a patient has expired, request information on the exact date of death, cause of death and if the patient expired at home/hospital.
  - a. Study staff will attempt to gather outcome information by inquiring whether the patient was re-hospitalized or had a medical visit for an infection prior to death.
  - b. A Medical Visit Reporting Form will also be completed.
- 2. Update the Physician Follow Up spreadsheet.
- 3. Patient will be added to the Trial Exit Report
- 4. The VTOC Enrollment survey will be updated.
  - a. Fill out Change of Enrollment Status section.
  - b. Enter Date of Death
  - c. Set Reason Disenrolled to "Death"
  - d. Add description under Notes for disenrolling.
- 5. Patient Tracking Log will be updated.
  - a. Highlight patient entry in red
  - b. Note "Patient deceased" and date of death in comments section

#### **Confirmed Lost to Follow Up:**

- 1. A patient will be considered confirmed lost to follow up when study staff are unable to contact patient for three or more months.
  - a. Contact attempts should include phone calls (to patient, alternate and emergency contacts), courtesy visit attempts, and engaging the original patient recruiter for new phone number/checking for readmission.
    - Central Office will:
- 2. Update the Physician Follow Up spreadsheet.
- 3. Add patient to the Trial Exit Report

- 4. Update VTOC Enrollment Survey
  - a. Fill out Change of Enrollment Status section.
  - b. Set Reason Disenrolled to "Lost to Follow Up".
  - c. Date Disenrolled is set to date of last known outcomes.
  - d. Add description under Notes for disenrolling.
- 5. Update Patient Tracking Log
  - a. Highlight patient entry in red
  - b. Note "Active disenrollment" and "Supervisor notified" in comments section

#### 10.11 Adverse Events

After receiving notification from a recruiter or patient via telephone/email that a study participant has experienced an adverse event, central office will:

- 1. Page study physicians using a secured intranet portal
- 2. A study physician will speak to patients who are reporting a study related AE.
- 3. Fill out Adverse Event Form on VTOC
  - a. Beneath "Unscheduled Events", click "New Record" next to "Adverse Event Reporting Form".
  - b. Fill out all information as possible according to the form.
- 4. Wait for the study physician's follow-up email & transcribe the assessments into the Physician Follow-Up spreadsheet:
  - a. Fill in information under tab marked "Adverse Events"
  - b. Save with current date.
- 5. The patient will be contacted by a study member daily until resolved (this will include any deemed non study related events) and updates will be entered into VTOC and Physician Follow-Up spreadsheet.

## 10.12 Medical Visit Reporting

If a patient indicates they have been to a hospital/NH/rehab center for any reason OR have visited the ER or outpatient clinic due to an infection, a Medical Visit Reporting Form must be completed and entered into VTOC.

- 1. To fill out Medical Visit Reporting Form on VTOC
  - a. Under "Unscheduled Events", click "New Record" next to "Medical Visit Reporting Form"





#### 10.13 Scanned Consents/Releases

All consent forms and HIPPA Authorization forms are to be filed electronically as well as within paper files as well. In order to ensure all consent forms are properly scanned, central office will:

- 1. Review Patient Tracking Log to see what consents need to be scanned.
  - a. "Y" for Yes will be placed in the corresponding cell to indicate that the consent signature page/surrogate signature form has been scanned.
- 2. Locate files in Central Office Cabinets
- 3. Create new folder w/ Study ID in the scanned consents folder
- 4. Go to "Xerox Scans" to find the newly scanned consents and rename each signature document.
  - a. Ex: D-2222-NL Consent or D-2222-NL Surrogate or D-2222-NL Release
- 5. Ensure consent is appropriately completed. If not, the study recruiter must be contacted immediately
- 6. Move renamed documents into appropriate folders
- 7. Open corresponding Consent without Signature Page
- 8. Append signature page
  - a. Go to Document  $\rightarrow$  Insert Pages  $\rightarrow$  From File
  - b. Select Patient's Consent Page (i.e. D-2222-NL) and insert at appropriate place
    - i. Double check after insertion that page numbers and consent versions match up
  - c. Save Document as Consent in the Scanned Consents folder (i.e. as D-2222-NL)

- i. You will be asked if you are sure you want to replace the current document
- ii. Click Yes

## 10.14 Creating Consent/Recruitment and Follow-Up Visit Packets

#### **Consent/Recruitment Packets:**

- \*Consent Packets should all have the following:
  - 1. Screening Form
  - 2. Consent Packet (Corresponding to hospital)
    - a. Consent Packets (UCI) to be used for UCI, Hoag or any post discharge recruitment.
    - b. Consent Packets (UCI) Spanish
    - c. Consent Packets (Mission)
    - d. Consent Packets (Memorial)
    - e. Consent Packets (Fountain Valley)
  - 3. Extra signature page (exempt Mission & Memorial) Spanish Signature Page
  - 4. HIPPA (UCI) Spanish HIPAA UCI
  - 5. HIPAA (Project CLEAR)- Spanish HIPAA Project Clear
  - 6. HIPAA (Memorial) only for Memorial Consents
  - 7. Contact Sheet Spanish Contact Sheet
  - 8. Enrollment Survey Spanish Enrollment Survey
  - 9. Medical Release Forms (2) Spanish Medical Release Forms (2)
  - 10. Consent Checklist Spanish Consent Checklist
  - 11. Dear Dr. Letter to be placed in the patient chart for the attending physicians

#### **Follow Up Visit Packets:**

- 1. Decolonization FU (English & Spanish)
  - a. Envelope for Cash
  - b. Cash Payment Form
  - c. Decolonization Follow-Up Survey (Spanish)
  - d. 2 Medical Visit Reporting Forms (Spanish)
  - e. 2 Adverse Event Forms (Spanish)
  - f. 2 Medical Visit Worksheets (Spanish)
- 2. Education FU (English & Spanish)
  - a. Envelope for Cash
  - b. Cash Payment Form
  - c. 2 Education Follow-Up Surveys (Spanish)
  - d. 2 Medical Visit Report Forms (Spanish)
  - e. 2 Medical Visit Worksheets (Spanish)

#### 10.15 PCP Letters

Primary Care Physician letters are generated for all patients.

#### 10.16 Exit Survey

The Trial Exit Survey should be conducted approximately one year after enrolled (i.e. 365 days after discharge or consent date, whichever is greater).

In order to complete the trial exit survey, central office will:

- 1. Check the Patient Tracking Log for Patients who are to complete their exit survey based on the above criteria.
- 2. Call patient and ask if he or she has a few minutes to complete a quick exit survey over the phone.
- 3. If so, Click on "New Record" underneath Exit Survey on VTOC.



- 4. Complete the questions listed within the trial exit survey
  - a. Fill out Medical Visit Form on VTOC if necessary (VTOC will prompt).
- 5. Thank the patient for participating in the trial.
- 6. Inquire if patient would be interested in future studies. Note their response in Communication Log, along with completion status of survey.
- 7. If a patient requests their lab results, inform the participant that the Senior Project Coordinator Supervisor will follow up within a week.
  - a. Each week, send Senior Project Coordinator Supervisor a list of patients who have requested their lab results.

## **10.17 Reports**

Central Office will distribute a study progress report to Senior Project Coordinator Supervisor and principal investigator daily. This progress report with include updates to the recruitment

numbers, dis-enrolled participants, follow up visits and status, as well as any other pertinent information involving the progress of the trial.

Additionally, quarterly reports will be sent to each participating facility's study champion and infection prevention team to inform them of the recruitment progress in the trial and at their site.

#### 10.18 Shipping

There will be situations where central office will assist with specimens that are shipped to UCI Medical Center for processing (from out of area visits or enrollment), as well as with the shipment of deidentified MRSA isolates that are sent to Rush University for resistance testing.

## 10.19 End of Day Laboratory Email

A summary email will be sent to the UCI microbiology lab daily to confirm the number of cultures that are to be received. A sample email is included below:



Recruitment visit bags include:

| Visit Type | Hibiclens | Bactroban | Periogard | Sponges | Container/Timer | Lotion | Pump |
|---|---|---|---|---|---|---|---|
| Recruitment | 1 | 3 | 1 | 3 | 1 | 1 | 1 |
| V1 | 1 | 4 | 1 | 4 | n/a | n/a | n/a |
| V2 | 2 | 6 | 2 | 6 | n/a | n/a | 1 |
| V3 | n/a | n/a | n/a | n/a | n/a | n/a | n/a |
| V4 | n/a | n/a | n/a | n/a | n/a | n/a | n/a |

## 11. Follow-Up Participant Tracking and Scheduling

Study personnel are responsible for keeping track of scheduled visits and updating contact information to ensure that subjects remain in the study. It is of the utmost importance that participant data are documented and kept well organized so as to avoid loss of information.

Harbor UCLA recruiters are responsible for following up with appointments for participants recruited from their facilities. UCI Central Office is responsible for following up on appointments for all other participants.

#### **UCI-based Enrollees**

Visit 1 appointments are scheduled by recruiters during the initial enrollment visit. Subsequent study visits (V2 – V4) are scheduled with the patient by the ICTS clinic nurse or coordinator/recruiter completing the follow up visits. UCI recruiters schedule appointments by calling the ICTS appointment line and then notifying UCI Central Office. ICTS nurses will record subsequent appointments into VTOC and email UCI Central Office on scheduled clinic visit dates, times and locations. UCI Central Office records all scheduled appointment into the Patient Tracking Log, ICTS appointment log or Recruiter appointment log, calendar, and ensures that the VTOC database is updated accordingly. Each Friday, UCI Central Office sends the ICTS nursing staff the appointment log to ensure that there are no discrepancies between the ICTS calendar and UCI Central Office records.

#### 11.1 Patient Contact

Contact information sheets for subjects will be kept in a locked cabinet when not in use. Contact information should be entered into VTOC within 24 hours of recruitment. All communication with a patient should be logged in the VTOC Communication Log. The date, time, mode, staff, urgency, category, and status in the Communication Log should be filled out along with the description of the communication with the patient.

UCI Central Office is responsible for tracking all important study events for UCI-based enrollees in the Patient Tracking Log excel spreadsheet and VTOC Communication Log. The log includes the patient Study ID, patient initials, recruiter initials, discharge date, decolonization plan (A/B),
clinic visit dates, decolonization regimen cycle start and end dates, and reminder phone call dates

### 11.2 Calendars

Subject scheduling will be managed through the study website calendar. Once a patient is enrolled, study coordinators are responsible for updating the calendar within 72 hours.

### 11.3 Call Lists

UCI uses the Patient Tracking Log to track which patients must be called for initial bathing, regular start bathing cycles, and appointment reminder calls. UCLA uses a similar tracking log to determine phone calls that must be made to patients. It is anticipated that VTOC will soon have a function to facilitate listing events such as bathing, appointments, and follow up that must be made on a given date or time period across all subjects in the VTOC database. Based on the event type and/or date enter as parameters, VTOC will list all patients requiring phone calls or additional follow back.

## 11.4 Patient Phone Calls

Patient phone calls are made by the UCI Central Office to the Decolonization patients up to five times per month. Patients assigned to the Decolonization group will be called after hospital discharge or on the date the patient indicated they would be able to start using the study products, the first and last day of their initial bathing cycle, the first day of their subsequent bathing cycles and the day prior to their scheduled clinic/home visits.

Patient phone calls are made by the UCI Central Office to the Education patients up to two times per month. Patients assigned to the Education group may be called after hospital discharge, on any day of the month to follow-up on any questions they may have regarding the educational materials and/or the study in general. Education patients will also be called the day prior to their scheduled clinic/home visits.

# 11.4.1 Initial Post-Discharge Phone Call

The UCI Central Office is responsible for calling each patient the next business day after hospital discharge. Patients assigned to the decolonization arm should be instructed to immediately begin their five day decolonization regimen. UCI Central Office will also answer any questions the patients might have about using the decolonization products or any general study questions. The toolkit binder should have been reviewed in full with each participant at the time of enrollment, so focused questions should be answered or a courtesy visit can be scheduled for additional support as requested by the participant.

Patients assigned to the Education Arm may also be called post-discharge, at the discretion of the recruiter, to answer any further questions about the study educational materials or any general study questions. The toolkit binder should have been reviewed in full with each participant at the

time of enrollment, so focused questions should be answered or a courtesy visit can be scheduled for additional support as requested by the participant.

### 11.4.2 Reminder Calls

Reminder phone calls for all study visits should be made 48 to 24 hours before the visit will occur. The outcome of reminder calls must be documented in the patient contact database. A message will be left if the subject does not answer. If a message cannot be left, coordinators will call the subject three times throughout the day. All phone call attempts will be documented in the patient contact database. Subjects will be called on 3 different days to attempt to reschedule the visit.

**Bathing:** Initial bathing (start & stop calls) - After PT has been discharged, each person (decolonization & education) is called to follow-up on the products given (binder/soaps & medicines), reinforce product start date adherence, answer general study questions and remind/ schedule V1.

**Monday calls**- All decolonization PTs are called on Mondays depending on Plan (A or B), see laminated calendar for assignment.

Decolonization patients have five day bathing cycles (Monday – Friday) twice a month. The dates of those cycles are determined on whether the patient is assigned to Plan A or Plan B.

### 11.4.3 Product Review/Orientation Calls

Project CLEAR. I was calling to see if you had any questions about the educational

materials or the products, and if you needed a refresher on how to use the products, I will

be in the area this Friday afternoon from 12-4. Please feel free to give us a call at



- 1. If the patients are education patients, the script will be modified to not reference the decolonization products.
- 2. If the patients are nursing home patients, the nursing home will be contacted by senior study staff for collaboration.

## 11.5 Study Helpline

A 1-800 helpline desk number plus an emergency pager number (the Senior Project Coordinator Supervisor) will be provided to the subjects. This 24-hour helpline is intended for Adverse Event reporting, urgent Medical Visit Reporting or any other urgent questions or concerns from study participants.

## 12. Bi-Monthly Phone Calls

Bi-monthly courtesy phone calls, intended to remind subjects of the upcoming study intervention, will occur the Friday prior to the 1<sup>st</sup> and 3<sup>rd</sup> or 2<sup>nd</sup> and 4<sup>th</sup> Monday of each month, depending on Plan A or Plan B. An additional call will be made on the Monday of a decolonization week to initiate the regimen and the Friday of a decolonization week to stop the intervention. A voicemail will be left if the subject does not answer. If voicemail is not available, coordinators will make three additional call attempts that day. All phone call attempts will be documented in the patient contact database.

Coordinators will call subjects who have been randomized to the intervention arm (serial decolonization) to:

- Remind them to begin the study intervention
- Inquire about adverse events
- Inquire about medical issues
- Re-educate patients on how to use the study products
- Answer any questions the subject may have

### **Start Regimen Script:**

"Hello, may I please speak to Mr. /Ms. <patient's last name>? My name is <caller's name> and I am calling from the Project CLEAR MRSA study to remind you to begin your five day Hibiclens bathing, nose ointment, and mouthwash regimen today. Will you be able to start today?"

(Patient says yes): "Great, the products work best against MRSA when you use all 3 together for all five days and don't miss any doses".

(Patient says no) – Find out why and if they can start the next day. If there is a delay in starting the regimen, be sure to have them start up as soon as possible and continue for five consecutive days.

"One last question for the study, we always ask that you let us know if you have been hospitalized for any reason or have had a clinic visit for a possible infection. Do you have either of those to report? Any other questions I can answer? Call us anytime toll free at

If the patient does not answer the call, it is acceptable to leave a message if the patient has indicated that messages may be left. Check the patient's contact sheet to see if they answered yes or no to "Is it okay to leave messages on this number?" Use the script below when leaving a message.

### **Start Regimen Message Script:**

"Hello Mr./Ms. <patient's last name>, I am calling from the Project CLEAR MRSA study to remind you to begin your five day Hibiclens bathing, nose ointment, and mouthwash regimen today. We also wanted to remind you to please let us know if you have been hospitalized for any reason or have had a clinic visit for a possible infection. We can be reached anytime toll free at \_\_\_\_\_\_\_."

Fill out a Medical Visit Reporting Form if a patient reports any hospitalizations for any reason or visits a clinic or doctor for a possible infection. Fill out an Adverse Event Reporting Form if the patient reports any adverse effects. See Section 14 for more information on reporting adverse events

### Add-on Lines to calls, rotating:

Scripted add-on to use when making calls/leaving messages (pick one or more & rotate):

- 1. Bactroban Since MRSA's main home is in the nose, be sure to use the nose ointment in the morning and at night during your 5-day bathing cycles to stop it from living in your nose.
- 2. Hibiclens Each time you bathe during your 5-day cycle, it is important to lather with the water off and leave the Hibiclens on your skin for 2 full minutes before rinsing off. It is also very important that you not use any other soaps, shampoos or lotions during your 5-day bathing cycles since some of them make Hibiclens stop working.
- 3. Periogard Sometimes MRSA will also live in the throat. Be sure to use the special mouthwash (Periogard) in the morning and at night during your 5-day cycles. Swish for 30 seconds and don't rinse with water immediately after using.
- 4. Your best chance of getting rid of MRSA is when you use all three products together. Let us know if you need more before your next visit with us.

The above statements can be followed with "Do you have any questions?"

#### **Additional Info:**

- ONLY stop bathing calls (prior to V3) when a patient requests not to be called.
  - Send email if possible to these patients.
- Any changes to PT's regimen Plan or to call list should be noted in Communication Log on VTOC and Patient Tracking Log.

## 13. Follow-up Study Visits

The UCI ICTS clinic hours for Project CLEAR are Mondays and Wednesday 8am-5pm at the UCI Medical Center in Orange, and Tuesdays and Thursdays 8am-5pm at the ICTS Clinic on the UC Irvine campus in Irvine. Weekends are available upon request.

The Harbor-UCLA CTRC Outpatient Clinic is open 7:30am to 4pm Monday through Friday. Subjects can be seen outside of these hours at the Inpatient CTRC Monday through Friday. Saturday follow-up visits can be arranged with prior notice.

Home and/or nursing home visits will occur when a subject is unable to come into the clinic for a study visit. Subjects who move or do not wish to have in-person visits may have their visit conducted over the telephone.

The follow-up visits occur at 1, 3, 6, and 9 months after the baseline visit.

Subjects will undergo the same body swabs as occur at the baseline visit and they will be administered a follow-up survey. Subjects will be compensated as outlined in Section 13.8.

# 13.1 Participant Education

If the participants request an additional patient education binder, it will be provided in their preferred language (English or Spanish).

Subjects will be provided reminder educational handouts specific to each follow-up visit. Study coordinators will review these handouts and any other information the subject would like to go over.

### 13.2 Interviews

The surveys will be completed in-person by study personnel. If the participant does not know or remember the answer, remind the participant to answer as best they can and move on the next question. The interview should take no more than 20 minutes.

### 13.3 Adverse Events

Adverse events will be recorded at the time the study coordinator becomes aware of the event. Study coordinators can be made aware of an adverse event in four ways:

- 1. The subject reports an event over the phone on a Bi-Monthly Call
- 2. The subject reports an event over the phone on a Reminder Call
- 3. The subject calls the 1-800 helpline number or pages the Senior Project Coordinator Supervisor
- 4. The subject reports an event at a follow-up visit

All adverse events will be followed until resolved, unless the subject exits the study and requests no contact.

Serious Adverse Events will be handled as described in the protocol Section 14.

### 13.4 Medical Events

If a patient affirms that they have been hospitalized or had an outpatient visit associated with a suspected MRSA infection on a phone call or follow-up visit, study coordinators will fill out a Medical Event Form and an Adverse Event Form with the subject. Patient will be asked to obtain records of their visit if easy to do so. Study coordinators will also contact the medical center the patient was seen at to request the medical records.

## 13.5 Body Site Swabbing

The same four body sites (nares, throat, groin/axilla, and wounds) will be swabbed at the follow-up visits. Refer to Section 9.5 for more information on how to swab body sites.

# 13.6 Scheduling Next Visit

Attempt to schedule the 1 month follow-up visit during the baseline visit whenever possible. If the participants cannot schedule the next visit, give them an appointment reminder card with the date on which the visit should occur. Two weeks before the 1 month follow-up visit, call the subject to schedule the appointment. The next study visit should always be scheduled at the current study visit; for example, the 6-month visit should be scheduled at the 3-month visit.

# **13.7 Update Contact Information**

Study coordinators must ask the subject to update their contact information prior to the end of all study visits. This includes:

• Phone number

- Address
- Emergency contact

## 13.8 Participant Payments

The participants will be compensated with cash at the completion of each follow-up visit.

- \$25 for the 1 month follow-up visit
- \$30 for the 3 month follow-up visit
- \$35 for the 6 month follow-up visit
- \$50 for the 9 month follow-up visit
- \$140 for the whole study

Fill out the Certification of Payment (see Figure 13.8) with the lead study coordinator's name, date, study IRB number, and the participant's name. Have the participant sign the receipt. At this time they will be given the cash.

Figure 13.8: Certification of Payment to Anonymous Persons – ICTS Irvine

| CERTIFICATION OF PAYMENT TO ANONYMOUS PERSONS - ICTS Irving 1. ADMINISTRATIVE INFORMATION | | | | | | | |
|---|---|---|---|---|---|---|---|
| | a. Contract/Grant to be charged: 9 - 445353 - 29070 - R - 03 - 3466 Loc Account Fund Project Sub Object Source | | | | | | |
| | b. Has a cash advance been issued? No Yes attach copy of check request | | | | | | |
| | c. IRB approval number or exempt registration number: | | | | | | |
| d. Principal Investigator Name: <u>Dr. Susan Huang</u> | | | | | | | |
| e. Department Unit Name: Project CLEAR-Changing Lives By Eradicating Antibiotic Resistance | | | | | | | |
| DISBURSEMENT CONTROL RECORD (please print) | | | | | | | |
| | Line | Date | Cash | Human | Paid To: Home Visits | | |
| | No. | Paid | V1-022<br>V2-020<br>V2-022 | Subject | | (Subject Signature) | Cash<br>Sign Out |
| | | | V0-000<br>V6-000 | ID Number | | IE<br>Sign Out 4 Home Visits | |
| | 1 | | | | | | |
| | 2 | | | | | | |
| | 3 | | | | | | |
| | 4 | | | | | | |
| | 5 | | | | | | |
| | 7 | | | | | | |
| | 8 | | | | | | |
| | 9 | | | | | | |
| | 10 | | | | | | |
| | Page | of | | Page Total | | | |
| | | | | Grand Total | | | |
| | | | | | | | 1 |
| 3. | I CERT | IFY THAT | THE AE | OVE INFORMAT | MON IS TRUE A | ND CORRECT. | |
| Principal (Co-Principal Investigator Date | | | | | | | |
| | | • | | | | | |
| Cev. 3/0 | 3 | | | | | | |

## 13.9 Off Site Follow-Up Visits

If the subject is unable to come in for the follow-up visit due to hospitalization or residence in a nursing home, study coordinators will complete the study visit at the medical center, nursing home, or patient's home, wherever the subject is currently residing.

### **13.9.1 Home Visit Procedures**

The following items are needed prior to the home visit:

- Project Clear Lab Coat (See VTOC for notes on patient preference for or against a lab coat)
- UCI Badge
- Gloves (Wear while swabbing patient)
- Anti-Bacterial gel/wipes
- Prepared Swabs (4 sterile swabs per bag with labels, carbon copy white/yellow form, and 1 white form)
- Pen
- Visit Compensation Amount (V1-\$25, V2-\$30, V3-\$35, V4-\$50) with small manila envelope
- "Certification of Payment to Anonymous Person ICTS Irvine" form (see Figure 13.8).
- Patients Name, ID Number, and Contact Details (address & directions)
- New Binder Sections:
  - V1: N/A
  - V2: "MRSA & Pets"
  - V2: General binder reminder
  - V3: V3 General binder reminder (Decol ONLY)
  - V4: N/A
- Calendar and area chart to book next visit (Month 1, 3, 6, 9)
- Staffed ICTS and Orange Clinic Visit Dates (Mon & Fri Orange; Tues & Thurs ICTS Irvine)
- Business card to write down next visit date and time for patient
- Pocket calendar note book or scrap paper to write next visit date to bring back to Central Office
- Trash Bag (for gloves, swab packaging, and to place empty Bactroban containers in after counting if Decolonization patient)

### If Patient is in Education Group:

- 1. "Participant Follow-up Survey Education"
- 2. "Medical Visit Reporting Form" x 2 (Same form used for Decolonization patient)

#### 3. "Medical Visit Worksheet" x2

### If Patient is in Decolonization Group:

- 1. "Participant Follow-up Survey Decolonization"
- 2. "Adverse Event Reporting Form" x 2
- 3. "Medical Visit Reporting Form" x 2 (Same form used for Education patient)
- 4. "Medical Visit Worksheet" x2
- 5. Prepackaged CHG Compliance Test Swabs (2 swabs per package with form)
- 6. Replenishment Products

### V1 Bags (1 month after enrollment)

- 1 Project Clear Canvas Bag (Containing below items)
- 4 Sponges
- 1 Hibiclens (1 bottle should last 2 months, ask how much used prior to visit)
- 4 Bactroban
- 1 Periogard
- 1 Pump (If needed)

### V2 Bags (3 months after enrollment)

- 2 x Project Clear Paper Bags
- 6 Sponges
- 2 Hibiclens (1 bottle should last 2 months, ask how much used prior to visit)
- 6 Bactroban
- 2 Periogard
- 1 Pump (If needed)

### Check Vision Tree (VTOC) for:

- Specific patient notes i.e. needs translator for patient or caregiver, non-communicative patients so look for the main contact, ability to be swabbed, unusual home conditions
- Notes on previous medical visits already recorded in VTOC so not duplicated

### Post Visit

- In VTOC, briefly report on visit in "Communication Log" (Ex: Home Visit (V1), completed.)
- Book Visit Date with Central Office. Enter next visit date on tracking log, VTOC, ENDMRSA calendar.
- Enter new survey data into VTOC. File hard copy into subject folder in locked cabinet. Ask Central Office for file cabinet key.
- Swabs to be transported to microbiology laboratory for processing
- If CHG compliance swabs were performed, bring back to office for logging and shipment preparation
- If adverse event form is completed email information as soon as possible to Central Office.
- Provide signed "Certification of Payment to Anonymous Person ICTS Irvine" to Central Office or sign back in money if visit was not completed with Fiscal Officer.

## 14. Adverse Event Reporting

Adverse events will be collected at the follow-up visits or when reported by the patient at any time. All adverse events should be inputted into the study database and the UCI CO should be notified immediately. The UCI CO will summarize the adverse event on the Adverse Event tracking log and will immediately notify the principal investigator of the adverse event. Adverse events reported for patients recruited from Harbor UCLA facilities should reported the Harbor-UCLA physician co-investigators. Adverse events reported for all other patients should be reported to the assigned study physician. The staff member completing adverse event should let the patient know that a study doctor will be following up with them.

Anticipated mild adverse events will be reported to the IRB on continuing review. All adverse events (mild and serious) will be summarized in the quarterly DSMB report. Serious Adverse Events (SAEs) requiring prompt reporting will be reported within the required timelines to the IRB and Data Safety and Monitoring Board. Any SAEs that result in a death must be reported to the UCI IRB and DSMB promptly, within 5 days.

## 15. Obtaining Medical Records

Complete medical records associated with the following will be requested from the appropriate medical center:

- The enrollment hospitalization
- Any subsequent hospitalization
- Any outpatient visit associated with any suspected infection, even if infection was not the purpose of the outpatient visit

All subjects will sign a page waiver allowing study personnel to request their medical records from any appropriate medical center. Study coordinators will fax, mail, or go in person to the request medical records as soon as the subject notifies them of the hospitalization or outpatient visit. If study coordinators do not receive the medical records within two weeks, they will send a repeat request up to 5 times. If incomplete records are received, another five attempts will be made to secure complete data.

# 16. Data Entry

Data entry will be performed by personnel at UCI and LA BioMed on a secure online database developed by Vision Tree Optimal Care (VTOC).

Figure 16.1: Vision Tree Optimal Care webpage.



All forms must be checked for completeness and accuracy before being entered by the data management team. Incomplete or inaccurate forms will be flagged and the responsible personnel will be contacted to verify answers on the form.

Inaccuracies will be recorded as a means of monitoring the quality of the data reported. Data quality reports will be issued monthly by the data management team.

## 17. Ordering Supplies

Each site will be responsible for ordering their own office and laboratory supplies.

The UCI group will be responsible for providing intervention toolkits and lab coats. UCI will also be responsible for emailing the latest versions of interviews, questionnaires, and other forms to the Project CLEAR Team.

The UCI group maintains a detailed inventory tracking log for all study supplies. Each item has an individual tracking sheet. Anytime a supply or product is taken from the central supply area, study personnel are responsible for recording the date, initials and number taken on the appropriate inventory sheet. UCI CO is responsible for monitoring inventory and requesting supplies before stock is depleted. When new stock is received, UCI CO updates the tracking log to reflect the number added

Decolonization supplies will be kept in a temperature controlled area.

# 18. Enrollment Reports

Enrollment reports that show the progress of recruitment are to be created daily and sent to the Principle Investigator and Senior Project Coordinator Supervisor each Friday. The report will be discussed each Monday at the investigative team call at 11:00 AM (PST). The enrollment report contains information about number of subjects enrolled per week and per month, progress by

recruiter and recruiting site, number exiting trial and distribution of participants by randomization scheme and study arm.

## 19. Specimen Delivery and Order Entry

Swab specimens collected from enrolled patients must be delivered to the appropriate microbiology laboratory within 24 hours of collection. Specimens collected from UCI associated facilities must be delivered to UCI Medical Center Microbiology laboratory at the end of each day. Specimens may also be dropped off at the Gottschalk Medical Plaza lab, before 5:00 pm, so that the courier service will transport the specimens to the UCI Medical Center Microbiology laboratory that same day.

The ICTS nurse or study coordinator/recruiter will fill out the Laboratory Requisition slip for the CLEAR Study Specimens for each patient. For the Laboratory Requisition slip the ICTS nurse or study coordinator/recruiter will be responsible for filling out the Subject ID, Collection Date, Specimen Collection Origin, Specimen Source and Visit. The ICTS nurse or study coordinator/recruiter will also be responsible for filling out his/her name, Date of Collection, Number Swabs Taken and Stamp the Study ID number in the four boxes to the left.

Study staff must notify UCI Central Office of all specimens they have collected for the day. UCI Central Office will record recruiter initials under Visited By, and log the Study ID, Visit Location, number of swabs, and Visit Type in the Central Office Lab Count Log. UCI Central Office will send the UCI Medical Center Microbiology laboratory an email (with cc: to UCI lead investigator and project supervisor) at the end of the day summarizing the specimens they should expect to receive for the day as shown in the table below.

| Visited By (Initials) | Study ID | <u>Visit Location</u> | # Swabs | Visit Type | <u>Recruiter</u> |
|---|---|---|---|---|---|

Visit number naming convention is R0 (initial recruitment), V1 (study visit 1), V2 (study visit 2), V3 (study visit 3), and V4 (study visit 4). The UCI Medical Center Microbiology laboratory sends a reply email verifying that all specimens are accounted for with the correct Study ID and paper work.

Should a problem arise the following is the contact information:

During regular hours – any issues, call or call after hours numbers if need assistance right away.

After hours, report of missing swabs etc..

The project assistant will bring the swabs to the lab. The bag with the specimens will be placed by the CLEAR assistant into the bin in the refrigerator in Central Processing. The bin will be marked CLEAR.

The swabs will be in a plastic bag clearly labeled PROJECT CLEAR containing a lab requisition form and CLEAR Specimen Sheet for each patient. The lab will place the specimen labels that

go with the corresponding patient on the CLEAR Specimen Sheet received. The Specimen Sheet will be kept in the lab and the lab requisition will be taken to Referral Services for billing.

The study location code CLR- will be documented in the medical record field.

Each swab will be labeled with the arm of the study (E or D), a study number (unique for each patient), and an alphabetical designation for randomization strata. The study-sample identifier will be entered into the patient name field during the specimen computer order-entry. In this way the specimen ID will appear on all labels. For example:

E1001, NN

This refers to E (education only group), 1001 is the patient identifier, NN means Non-Hispanic/Non-long term care facility.